CLINICAL TRIAL: NCT05548582
Title: A Randomized Controlled Trial to Study Reduced Opioid Prescription After Laparoscopic Hysterectomy
Brief Title: Reduced Opioid Prescription After Laparoscopic Hysterectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00345074
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pain, Postoperative; Opioid Misuse; Opioid Use; Pain
MeSH Terms: conditions — Pain, Postoperative; Opioid-Related Disorders; Pain | interventions — Oxycodone; Tablets; Acetaminophen; Ibuprofen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-operative opioid prescription (Other): Ibuprofen 600mg every 6 hours x 48 hours then as needed (total 30 tablets). If allergy or contraindication to ibuprofen, then will receive Meloxicam 15mg daily x 48 hours then as needed
  Acetaminophen 500mg every 6 hours x 48 hours then as needed (total 30 tablets)
  Oxycodone 5mg every 4 hours as needed (total 12 tablets)
  Interventions: Drug: OxyCODONE 5 mg Oral Tablet; Drug: Acetaminophen 500 mg Tab; Drug: Ibuprofen 600 mg
- No Opioid prescription (Active Comparator): Ibuprofen 600mg every 6 hours x 48 hours then as needed (total 30 tablets). If allergy or contraindication to ibuprofen, will receive Meloxicam 15mg daily x 48 hours then as needed
  Acetaminophen 500mg every 6 hours x 48 hours then as needed (total 30 tablets)
  Interventions: Drug: Acetaminophen 500 mg Tab; Drug: Ibuprofen 600 mg

INTERVENTIONS:
Drug: OxyCODONE 5 mg Oral Tablet — No opioid prescription after laparoscopic hysterectomy
  Arms: Post-operative opioid prescription
Drug: Acetaminophen 500 mg Tab — Standard prescription
Drug: Ibuprofen 600 mg — Standard prescription

SUMMARY:
Given the nationwide epidemic of opioid use and abuse (in part due to over prescription), this study aims at addressing the need for opioid prescription after laparoscopic hysterectomy.

DETAILED DESCRIPTION:
Currently, there is a nationwide epidemic of opioid abuse and overdose deaths. One source of excess opioids is overprescribing in the postoperative period. Given the increasing opioid abuse and over-prescription post-operatively, an effort must be made to determine whether non-opioid multimodal medications are adequate in treating postoperative pain after laparoscopic hysterectomy and would not increase the need for additional prescriptions or unscheduled patient contacts. This study aims to find the optimal prescriptions for pain after laparoscopic hysterectomy in an attempt to eliminate opioid use.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 undergoing outpatient laparoscopic (conventional or robotic) hysterectomy for benign indications

Exclusion Criteria:

* Allergy or other contraindication to the prescribed medications such as acetaminophen, ibuprofen, or oxycodone
* Known opioid use or abuse (defined as reported use or treatment for abuse within the last 3 months)
* Chronic pain patients
* Conversion to laparotomy
* Malignancy as the indication for surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score on post-operative day one | 1 day
  Numeric pain score on post-operative day one: patient reported pain using the Likert pain scale from 0 to 10
Pain score on post-operative day seven | 7 days
  Numeric pain score on post-operative day seven: patient reported pain using the Likert pain scale from 0 to 10

SECONDARY OUTCOMES:
Satisfaction of pain control on postoperative day one | 1 day
  Overall satisfaction of pain control on postoperative day one (binary question - Yes/No)
Satisfaction of pain control on postoperative day seven | 7 days
  Overall satisfaction of pain control on postoperative day seven (binary question - Yes/No)
Mobility on postoperative day one | 1 day
  Satisfaction with mobility on postoperative day one (binary question - Yes/No)
Mobility on postoperative day seven | 7 days
  Satisfaction with mobility on postoperative day seven (binary question - Yes/No)
Total opioid consumption on postoperative day one | 1 day
  Total narcotic consumption by postoperative day one (in morphine milligram equivalent)
Total opioid consumption on postoperative day seven | 7 days
  Total narcotic consumption by postoperative day seven (in morphine milligram equivalent)
Opioid related side effects on postoperative day one | 1 day
  Presence of opioid related side effects such as nausea, vomiting, constipation, dizziness, abdominal distention, and itchiness on postoperative day one (binary question - Yes/No)
Opioid related side effects on postoperative day seven | 7 days
  Presence of opioid related side effects such as nausea, vomiting, constipation, dizziness, abdominal distention, and itchiness on postoperative day seven (binary question - Yes/No)
Unplanned calls/visits | 7 days
  Unplanned visits to the emergency room or clinic and unexpected patient initiated phone call related to pain control postoperatively (binary question - Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Borahay, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States